CLINICAL TRIAL: NCT04570709
Title: Feasibility and Acceptability of A RN-Led Palliative and Supportive Care Intervention for Adults With Acute Leukemia
Brief Title: RN-Led Palliative and Supportive Care Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC1848; 5R34NR019131 (NIH)
Record Dates: First submitted 2020-02-11; First posted 2020-09-30 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Symptoms; Function; Quality of life; Acute myeloid leukemia; Palliative care; Supportive care
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This is a feasibility study. This study is conducted on one unit and to reduce bias and contamination, the control patients will be recruited and consented first. After recruitment of the 20 control patients, we will then recruit 20 intervention patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in the control arm will receive standard of care and no intervention.
- Intervention (Experimental): Patients in the intervention arm will receive the PACT intervention provided by a multidisciplinary team of RNs, OTs, and PTs.
  Interventions: Other: Palliative And supportive Care inTervention (PACT)

INTERVENTIONS:
Other: Palliative And supportive Care inTervention (PACT) — Using the Adaptive Leadership Framework for Chronic Illness as a guide. The nurse, occupational and physical therapists will meet with the patient and caregiver after the baseline assessment to discuss their Specific, Measurable, Achievable, Relevant, and Time-Bound (SMART) goals. Additionally, the occupational and physical therapists will provide the patient a PACT intervention binder. Regular phone calls or visits from a registered nurse, occupational therapists, and physical therapists for patients and caregivers in the intervention.
  Arms: Intervention

SUMMARY:
This single institution feasibility and acceptability study includes patients with acute leukemia which is designed to examine a novel palliative and supportive care intervention (Palliative and supportive Care inTervention; PACT) in which registered nurses (RNs), occupational therapists (OTs), and physical therapists (PTs) address the activity needs of older adults with acute leukemia during their hospital stay.

DETAILED DESCRIPTION:
The primary objective of the study is to assess feasibility, acceptability, and change in pre and post measures of symptoms, function, and QOL by administering the PACT intervention. The first 20 participants in the control group will receive usual care. The next 20 participants will receive the PACT intervention. Each participant in the intervention group will be cared by a collaborative, multidisciplinary, integrated team including RNs, OTs and PTs.

ELIGIBILITY:
[Patient]

Inclusion Criteria:

1. ≧60 years of age
2. Diagnosis of acute myeloid leukemia
3. Receive low-dose cytarabine or hypomethylating agent (HMA) in combination with Venetoclax chemotherapy
4. Speak and read English
5. Preference will be given to patients with care partners

Exclusion Criteria:

1. Patients receiving hospice care

[Caregiver]

Inclusion Criteria:

1. ≧18 years of age
2. Identified by patient as caregiver
3. Speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2024-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Bryant, PhD, RN, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Lineberger Comprehenisive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 09/14/2020 through 04/06/2023 at one cancer center in North Carolina. Subjects were enrolled in the study between 09/14/2020 - 4/4/2023.
Pre-assignment Details: A total of seventy-two participants consented to the study, but five of them withdrew their consent during screening and therefore were not enrolled in the study.
Groups:
- Intervention: Patients in the intervention arm will receive the PACT intervention.
- Care Partner -Control: Subjects who are family or friends or support patients in the control group
- Care Partner- Interventional: Subjects who are family or friends or support patients in the intervention group.
Period: Overall Study
Arm/Group | Control | Intervention | Care Partner -Control | Care Partner- Interventional
Started | 20 | 18 | 14 | 15
Completed | 20 | 18 | 14 | 13
Not Completed | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Subjects who were joined to the study. Care Partner -Control" and "Care Partner- Interventional" Arms were not assessed for this Baseline Measure support person and miles traveled to the clinic.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Care Partner -Control | Care Partner- Interventional | Total
Number analyzed (Participants) | 20 | 18 | 14 | 15 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.7 (7.49) | 74 (6.75) | 65.6 (9.3) | 67.4 (13.12) | 70.43 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 13 | 12 | 53
  Male | 5 | 5 | 1 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 20 | 14 | 12 | 14 | 60
  Unknown or Not Reported | 0 | 3 | 2 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 1 | 3
  Black or African American | 1 | 3 | 1 | 3 | 8
  White | 17 | 13 | 13 | 11 | 54
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 14 | 15 | 67
Education [Count of Participants; unit: Participants]
  1st-8th grade | 0 | 2 | 0 | 0 | 2
  9-11th grade | 0 | 0 | 1 | 2 | 3
  High school graduate/GED | 9 | 5 | 3 | 7 | 24
  College Degree | 4 | 10 | 6 | 5 | 25
  Advanced Degree | 6 | 1 | 4 | 1 | 12
  Prefer not to answer | 1 | 0 | 0 | 0 | 1
Marital Status [Count of Participants; unit: Participants]
  Single, never married | 0 | 0 | 1 | 0 | 1
  Married/partnered | 14 | 14 | 12 | 14 | 54
  Divorced | 3 | 2 | 1 | 1 | 7
  separated | 0 | 1 | 0 | 0 | 1
  widowed | 3 | 1 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Acceptability
Description: Feasibility and acceptability will be assessed as the number of participants who were approached, consented to, and eligible for the study.
Time Frame: Baseline
Population: Potential research participants screened.
Measure: Count of Participants; unit: Participants
Groups:
- Potential - Eligible- Consented Participants: The number of subjects who were approached, eligible and consented.
Arm/Group | Potential - Eligible- Consented Participants
Number analyzed (Participants) | 128
Participants
  Screened | 128
  Eligible | 93
  Approached | 54
  Consented | 38

2. Primary Outcome: Retention Rate
Description: The rate of participants who consented to the study completed study intervention at the time point.
Time Frame: Baseline and up to 30 days (first and second cycles)
Population: Subjects started the study and completed the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 20 | 18
Participants
  Consented | 20 | 18
  Cycle 1 | 20 | 18
  Cycle 2 | 15 | 15

3. Primary Outcome: Symptom Monitoring Data Collection Rate
Description: The number of participants who joined the study and symptom monitoring were assessed at the time point.
Time Frame: Baseline and up to 30 days (first and second cycles)
Population: Subjects started the study and were assessed at the time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 20 | 18
Participants
  Cycle 1 | 17 | 12
  Cycle 2 | 14 | 10

4. Primary Outcome: Caregiver Follow-Up Data Collection Rate
Description: Caregiver Follow-Up data collection rate was assessed the number of caregiver participants who joined the study and symptom monitoring was assessed at the time points.
Time Frame: At second cycle (at days 30)
Population: Caregivers of subjects started the study and responded the questions at the time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Care Partner -Control | Care Partner- Interventional
Number analyzed (Participants) | 14 | 15
Participants | 10 | 12

5. Primary Outcome: Comparison of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score in Cycle 1.
Description: Mean Overall, Physical, Emotional, and Fatigue Quality of Life (QOL) scores were assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) in control and intervention arms at Cycle 1.
  The EORTC QLQ-C30 is a cancer-specific instrument with 30 questions that incorporates 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 9 symptom scales (fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties); and a global health and quality-of-life scale. Most questions used a 4-point scale (1 =Not at all to 4 =Very much); 2 questions used a 7-point scale (1 =Very poor to 7 =Excellent). A higher score=better level of functioning or greater degree of symptoms. The scores of these scales were averaged from the scores of the component items, transformed, and analyzed on a 0 - 100 scale.
Time Frame: Baseline, up to 30 days
Population: Subjects who were joined to the study and completed assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 20 | 18
score on a scale
  Cycle1 Overall QoL | 55.8 (22.6) | 52.8 (25.7)
  Cycle1 Physical QoL | 72.3 (22.6) | 64.4 (27.7)
  Cycle1 Emotional QoL | 83.3 (15.3) | 77.3 (22.3)
  Cycle1 Fatigue | 49.4 (29.8) | 53.1 (30.1)

6. Primary Outcome: Comparison of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score in Cycle 2.
Description: Mean Overall, Physical, Emotional, and Fatigue Quality of Life (QOL) scores were assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) in control and intervention arms at Cycle 2.
  The EORTC QLQ-C30 is a cancer-specific instrument with 30 questions that incorporates 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 9 symptom scales (fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties); and a global health and quality-of-life scale. Most questions used a 4-point scale (1 =Not at all to 4 =Very much); 2 questions used a 7-point scale (1 =Very poor to 7 =Excellent). A higher score=better level of functioning or greater degree of symptoms. The scores of these scales were averaged from the scores of the component items, transformed, and analyzed on a 0 - 100 scale.
Time Frame: 30 days after starting to the study
Population: Subjects who were joined to the study and completed the assessment on Cycle 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 15 | 15
score on a scale
  Cycle2 Overall QoL | 64.4 (16.8) | 60.1 (20.5)
  Cycle2 Physical QoL | 76.9 (18.0) | 72.9 (19.8)
  Cycle2 Emotional QoL | 86.7 (10.8) | 87.5 (15.6)
  Cycle2 Fatigue | 39.3 (17.2) | 54.0 (30.5)

7. Primary Outcome: Comparison of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Scores Between Cycle 1 and Cycle 2.
Description: Overall, Physical, Emotional, and Fatigue Quality of Life (QOL) scores were assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) in the intervention arm both at Cycle 1 and 2. Score difference for each subject and mean differences between scores were calculated.
  The EORTC QLQ-C30 is a cancer-specific instrument with 30 questions that incorporates 9 multi-item scales. Most questions used a 4-point scale (1 =Not at all to 4 =Very much); 2 questions used a 7-point scale (1 =Very poor to 7 =Excellent). A higher score=better level of functioning or greater degree of symptoms. The scores of these scales were averaged from the scores of the component items, transformed, and analyzed on a 0 - 100 scale.
Time Frame: Baseline and until day 30 (Cycle 1 and Cycle 2)
Population: Subjects who were joined to the study and responded to (EORTC QLQ-C30) questionnaire at Cycle 1 and Cycle 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Group: Patients in the intervention arm will receive the PACT intervention assessed in both Cycle 1 and Cycle 2.
Arm/Group | Intervention Group
Number analyzed (Participants) | 14
score on a scale
  Overall QOL | 5.36 (26.27)
  Physical QOL | 3.81 (24.35)
  Emotional QOL | 7.34 (13.66)
  Fatigue | 4.76 (33.39)

8. Primary Outcome: Treatment-related Symptoms as Assessed by Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: 19 items include diarrhea, chills, heartburn, nausea, appetite, mouth sores, vomiting, constipation, cough, rash, shortness of breath, fatigue, anxiety, sadness, nothing will cheer me up, pain, insomnia, concentration, and memory. The severity is assessed from "None" to "Very severe" and the interference level is assessed from "Not at all" to "Very much."
Time Frame: Up to180 days
Population: Subjects started the study and responded to the PRO-CTCAE questionnaire at the time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 20 | 18
Participants
  diarrhea | 9 | 13
  chills | 12 | 15
  heartburn | 7 | 13
  nausea | 8 | 14
  appetite | 11 | 15
  mouth sores | 8 | 15
  vomiting | 1 | 9
  constipation | 10 | 15
  cough | 8 | 15
  rash | 3 | 0
  shortness of breath | 9 | 15
  fatigue | 12 | 15
  anxiety | 9 | 14
  sadness | 8 | 14
  nothing will cheer me up | 7 | 11
  pain | 8 | 8
  insomnia | 11 | 15
  concentration | 10 | 14
  memory | 10 | 14

ADVERSE EVENTS:
Description: The protocol does not require Adverse Event Collections and/or All-Cause Mortality data. Deaths and adverse events were not assessed.
Arm/Group | Control | Intervention | Care Partner -Control | Care Partner- Interventional
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04570709/Prot_SAP_000.pdf